CLINICAL TRIAL: NCT05017506
Title: Turkish Validity and Reliability Study of The Coronavirus Impact Scale
Brief Title: The Coronavirus Impact Scale Validity and Reliability Study
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Assoc. Dr., Ordu University
Other Study IDs: ayyuzlum3207*
Record Dates: First submitted 2021-08-16; First posted 2021-08-24 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: TURKISH VALIDITY AND RELIABILITY STUDY OF THE CORONAVIRUS IMPACT SCALE
Keywords: Coronovirus, Impact, Reliability, Validity, Measuring tool, Nursing.
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A survey will be made. — A survey will be made.

SUMMARY:
This research; The Turkish validity and reliability study of the "Coronavirus Impact Scale" developed by Stoddard and Kaufman (2020) will be conducted in order to bring a new measurement tool to our country.

DETAILED DESCRIPTION:
This research; The Turkish validity and reliability study of the "Coronavirus Impact Scale" developed by Stoddard and Kaufman (2020) will be conducted in order to bring a new measurement tool to our country.

Method: This research was planned as a methodological study. Research Question: Is the "Coronavirus Impact Scale" a valid and reliable measurement tool for Turkish society?

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old,
* At least primary school graduate,
* Able to communicate verbally and
* Persons who agree to participate in the research will be included in the research.

Exclusion Criteria:

* Psychiatric illness and unable to communicate,
* Having a language problem
* Persons who do not have the skills to read and understand the questionnaire will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults presenting to outpatient clinics in the hospital.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Coronavirus Impact Scale | 8 months
  The Coronovirus Impact Scale was developed by Stoddard and Kaufman (2020) to assess the impact of Covid-19 on people. The scale consists of 12 questions. Questions 1-9 in the scale are in 4-point Likert type, 0. There is no change, 1. Mild, 2. Moderate and 3. Severe, and points are taken between 0-3 from these questions. The questions between 10 and 11 on the scale are in a 5-point Likert type and are scored between 0-4 (indicating that from mild symptoms to death). However, the number of first degree family members diagnosed with coronavirus in question 10 and the number of relatives or close friends diagnosed with coronavirus in question 11 are not taken into account in the scale. The 12th question of the scale is open-ended and determines the other aspects that the coronavirus epidemic affects life. A minimum score of 0 and a maximum score of 35 are obtained from the scale, and as the score increases, the degree of exposure of people to the Corona virus increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu Univercity, Ordu, Cumhurıyet Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz Yavuz A, Altinsoy C, Toraman MN, Karabulut Musdal N. The Turkish validity and reliability of the Reward-Based Eating Drive (RED-13) Scale. PLoS One. 2025 Apr 25;20(4):e0322097. doi: 10.1371/journal.pone.0322097. eCollection 2025. PMID 40279302
- See also: Stoddard J, Kaufman J. (2020). Coronavirus Impact Scale. — https://www.phenxtoolkit.org/toolkit_content/PDF/CIS_Stoddard.pdf